CLINICAL TRIAL: NCT00803335
Title: The Effects of Local Vaginal Estrogen in Postmenopausal Women With Pelvic Organ Prolapse: A Randomized Control Trial
Brief Title: The Effects of Local Vaginal Estrogen in Postmenopausal Women With Pelvic Organ Prolapse
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 08135-08-076
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2014-02

CONDITIONS: Pelvic Organ Prolapse; Vaginal Atrophy
Keywords: pelvic organ prolapse; vaginal atrophy; atrophic vaginitis; postmenopausal; posthysterectomy; vaginal health; vaginal cytology; vaginal maturity index; vaginal histology; quality of life questionnaires
MeSH Terms: conditions — Pelvic Organ Prolapse; Atrophic Vaginitis | interventions — Estrogens, Conjugated (USP)

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Premarin cream 0.5gm (Active Comparator): Application of 0.5gm of vaginal estrogen cream nightly until surgery.
  Interventions: Drug: Vaginal conjugated estrogen cream 0.5gm
- Premarin cream 1.0gm (Active Comparator): Application of 1.0gm of vaginal estrogen cream nightly until surgery.
  Interventions: Drug: Vaginal conjugated estrogen cream 1.0gm
- No intervention (No Intervention): Women in this arm will not apply any cream or moisturizers to the vagina until surgery, ie no intervention.

INTERVENTIONS:
Drug: Vaginal conjugated estrogen cream 0.5gm — Women in this arm will apply 0.5gm vaginal estrogen cream nightly until surgery.
  Other Names: Premarin
  Arms: Premarin cream 0.5gm
Drug: Vaginal conjugated estrogen cream 1.0gm — Women in this arm will apply 1.0gm vaginal estrogen cream nightly until surgery.
  Other Names: Premarin
  Arms: Premarin cream 1.0gm

SUMMARY:
The purpose of this study is to find out how long it takes the vagina to respond to hormonal vaginal cream in women with pelvic organ prolapse (bulge in the vagina). It also will address the appropriate amount to use prior to vaginal repair of pelvic organ prolapse.

DETAILED DESCRIPTION:
Subjective and objective vaginal health symptoms, validated pelvic floor questionnaires, cytology and histology will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 45 years or older
* Postmenopausal (>55 if natural menopause)
* Clinical atrophic vaginitis (at least mild atrophy)
* Pelvic organ prolapse(at least stage 2 or greater)
* Posthysterectomy
* Surgery date between 2-12 weeks after recruitment

Exclusion Criteria:

* Uterus present
* Well-estrogenized appearing vagina
* Known or suspected history of breast carcinoma
* Hormone-dependent tumor
* Genital bleeding of unknown cause
* Acute thrombophlebitis or thromboembolic disorder associated with estrogen use
* Vaginal infection requiring treatment
* Allergy to estrogen or its constituents
* Any serious disease or chronic condition that would interfere with study compliance or preoperative surgical clearance.
* Use of exogenous corticosteroid or sex hormones (including homeopathic preparation) within the 8 weeks prior to recruitment
* Initiation or continuation of anticholinergic medication (which could bias the results of the pelvic floor questionnaires)

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2008-12; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Vaginal tissue samples obtained at the time of vaginal repair of pelvic organ prolapse will be analyzed for epithelial and subepithelial thickness, vascularity and inflammatory cells using standard H&E stains. | baseline and 2-12 weeks after treatment (at time of surgery)

SECONDARY OUTCOMES:
Vaginal histology will be compared to validated pelvic floor quality of life questionnaires, vaginal health symptoms, vaginal health scoring, and vaginal cytology. | baseline and 2-12 weeks after treatment (at time of surgery)

CONTACTS AND LOCATIONS:
Overall Officials: Christine M Vaccaro, DO, Principal Investigator — Good Samaritan Hospital
Locations (1):
- Trihealth (Good Samaritan Hospital, Bethesda North Hospital), Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Taithongchai A, Johnson EE, Ismail SI, Barron-Millar E, Kernohan A, Thakar R. Oestrogen therapy for treating pelvic organ prolapse in postmenopausal women. Cochrane Database Syst Rev. 2023 Jul 11;7(7):CD014592. doi: 10.1002/14651858.CD014592.pub2. PMID 37431855